CLINICAL TRIAL: NCT00453609
Title: Injectable Naltrexone Treatment of Alcohol Dependence in Serious Mental Illness (SMI): An Open Prospective Pilot Trial
Brief Title: Injectable Naltrexone Treatment of Alcohol Dependence in Serious Mental Illness (SMI)
Acronym: vivitrol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUNY Upstate MU IRB # 5463
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Alcohol Dependence
Keywords: Bipolar Disorders; Schizophrenia; Schizoaffective Disorders; Alcohol Dependence; Long-lasting injectable naltrexone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: long-lasting injectable naltrexone

SUMMARY:
The overall goal of this project is to improve the treatment of alcohol dependence in patients with serious mental illness (SMI). SMI for this study is defined as any patient with any of the following diagnoses: schizophrenia, schizoaffective disorder, and bipolar type I or type II disorder. Alcohol and other substance use disorders (SUDs) are common among individuals with SMI. SUD comorbidity is associated with many adverse consequences. However, to date, few reports have addressed the efficacy of pharmacological treatments for SUDs in this population. Naltrexone pharmacotherapy is an effective treatment for alcohol dependence, but it has not been systematically applied to the care of patients with SMI. The primary aim of this study is to determine the feasibility of long-acting injectable naltrexone administration in a clinical trial in patients with SMI who also have a diagnosis of alcohol dependence. Secondary aims include providing a preliminary assessment of the tolerability and safety of long-acting injectable naltrexone in patients with SMI who also have a diagnosis of alcohol dependence. An additional aim is to provide a preliminary assessment of the efficacy of long-acting injectable naltrexone in reducing alcohol use from baseline levels.

DETAILED DESCRIPTION:
The proposed project is a 1-year pilot program of research, which will examine the feasibility of a new, intramuscular (IM) long-acting form of naltrexone. The long-acting form of naltrexone may improve medication adherence, which has been shown to be critical to successful naltrexone treatment of alcohol dependence. The study is a 16-week, randomized, prospective, open-label trial, including a 12-week course of monthly naltrexone injections. A follow-up interview will be conducted 4 weeks after discontinuation of medication. Thirty subjects will be recruited. Voucher-based incentives will be provided to all subjects to ensure attendance for medication administration. Weekly motivational counseling sessions will be conducted and will focus on improving motivation to stop alcohol use. Study outcomes consist of self-report and biological measures of alcohol use; measures of psychiatric symptom severity and neurocognitive functioning; and genetic testing to examine functional polymorphism (Asn40Asp) differences in the subjects' μ-opioid receptors (OPRM1), which may predict response to naltrexone treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 to 69, with a DSM-IV diagnosis of Schizophrenia, Schizoaffective Disorder, or Bipolar Type I or Type II Disorder.
2. DSM-IV diagnosis of Alcohol Dependence in the last 12 months.
3. Level of Drinking:

   1. At least four days of drinking in the 30 days prior to consent and/or during screening period OR
   2. For prospective subjects who are currently in an inpatient or residential facility or recently discharged within 30 days prior to consent: At least 4 days of drinking during the period of time immediately prior to inpatient admission and/or during post-discharge.
4. Currently prescribed antipsychotic medications, mood stabilizers, or antidepressants.
5. One negative urine screen for opiates prior to start of medication and a self-report of no opioid use for at least 1 week prior to starting medication.
6. Currently involved in outpatient psychiatric treatment at one of the study sites (Hutchings Psychiatric Center, SUNY Upstate Adult Psychiatric Clinic, St. Joseph's Hospital, VA Medical Center) or at another location in the community.

Exclusion Criteria:

1. Inability to give adequate informed consent;
2. Currently taking disulfiram (Antabuse), naltrexone, or acamprosate (Campral);
3. Current DSM-IV diagnosis of Opioid Dependence (criteria met in the last month);
4. Current regular use of prescribed opioid analgesics, such as methadone, morphine, codeine, meperidine, and all other opioids. If the subject reports taking a prescribed opioid analgesic only occasionally, the study physician or nurse practitioner will contact the prescribing physician regarding the safety of study participation and the possibility of using an alternative. The principal investigator will make the final determination after obtaining the primary physician's recommendation regarding this criterion.
5. Current daily use of non-prescribed opioids.
6. Currently taking ibuprofen or other potentially hepatotoxic medications in amount and/or frequency judged by the Principal Investigator to pose clinically significant added risk of hepatic injury;
7. Female patients of childbearing potential who are sexually active, not sterile, and who deny using birth control;
8. Female patients who are pregnant or nursing;
9. Significant unstable medical problems, including any significant unstable psychiatric disorders. The study physician conducting the medical history and physical exam will exclude such clinically unstable individuals;
10. AST (aspartate aminotransferase test) levels: If AST is greater than 3x upper limit of normal;
11. Subjects who do not attend required screening appointments. Subsequent exclusion from the study for reasons related to non-attendance will be based on the judgment of the principal investigator;
12. In need of acute medical detoxification from alcohol in the judgment of the study physician based on results a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale Based on DSM-III-R (CIWA-AD) and other information obtained;
13. Scheduled surgery within 3 months of intake;
14. Subjects who have pending legal proceedings whose outcome may lead to incarceration within 3 months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
feasibility: number recruited, visits attended

SECONDARY OUTCOMES:
genetic testing to examine functional polymorphism (Asn40Asp) differences in the subjects' μ-opioid receptors (OPRM1)
alcohol use: self-report, biological measures, level of craving.
psychiatric functioning
neuropsychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Batki, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (3):
- United States (3):
  - St. Joseph's Mental Health Services, Syracuse, New York
  - Hutchings Psychiatric Center, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York

REFERENCES:
- See also: SUNY Upstate Medical University — http://www.upstate.edu/